CLINICAL TRIAL: NCT01206621
Title: Assessment of the Utility of Vibration Response Imaging (VRI) in Evaluating Dyspnea Patients Presenting to the Emergency Department
Brief Title: Vibration Response Imaging (VRI) in Dyspnea Patients Presenting to the ED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deep Breeze (Industry)
Responsible Party: Merav Gat, VP of Clinical & Regulatory Affairs, Deep Breeze
Other Study IDs: DB051
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2010-09

CONDITIONS: Dyspnea
Keywords: dyspnea; COPD; CHF; asthma
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood drawn for BNP testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED patients presenting with dyspnea

SUMMARY:
For the patient with acute dyspnea in the ED, early differentiation between CHF and non-CHF causes is essential for proper management. The capacity to triage patients quickly and accurately has a beneficial impact upon outcome, disposition, stratification and length of stay in the ED and required length of hospital admission.

The ability to assess pulmonary status rapidly by quantitative regional vibration technology offers significant potential advantage for earlier diagnosis. The VRI technique may provide a quick and accurate method of differentiating between dyspnea due to HF and dyspnea due to pulmonary causes; thereby improving management and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide Informed Consent;

  ->40 years of age;
* Estimated Body Mass Index >19;
* Patient presented to the emergency department with a chief complaint of acute dyspnea.

Exclusion Criteria:

* Patients with obvious trauma or acute anxiety as a cause of dyspnea;
* Patient has already received directed therapy in the ED and symptoms are remarkably improved;
* Physician concern regarding possible harm to patient caused by positioning or ambulating the patient for VRI testing;
* Intubated or mechanically ventilated;
* Acute hemodynamic or ventilator instability requiring immediate resuscitation;
* Body habitus or skin condition that might prevent the placement of the sound sensors on the back (e.g. severe scoliosis, kyphosis, chest wall deformation, skin lesion on the back or compression fracture);
* Hirsutism.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED with acute dyspnea who are greater than 40 years of age and consisting of both male and females
Sampling Method: Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Assess the ability of the VRI to improve clinical outcomes via accurate, early classification of the cause of acute dyspnea as HF or other (i.e. COPD, PE etc). | Baseline testing at ED presentation
  The primary efficacy analysis set (PEAS) consists of all patients who have Gold Standard (GS) diagnosis (CHF/non-CHF) & VRI records.
  * Accuracy rate is defined as the accuracy between the GS and VRI.
  * Accuracy parameters between the GS and VRI will be calculated using accuracy rate, sensitivity, specificity, negative predictive value (NPV), positive predictive value (PPV) & likelihood ratios (+,-).

SECONDARY OUTCOMES:
Assess the agreement to aid in classifying the cause of acute dyspnea as HF or other of the VRI in comparison to BNP/NTproBNP assays. | Baseline testing at ED presentation
  The secondary efficacy analysis set (SEAS) consists of all patients who have final diagnosis (CHF/non-CHF), BNP/NT-proBNP & VRI results.
  * Agreement rate (2X2 agreement table) between BNP/NT-proBNP (based on separate decision cut-offs for each assay) and VRI will be calculated for dyspnea due to CHF or other causes.
  * The discordant observations (from the agreement table) will be further evaluated between the VRI and GS.
  * Logistic regression will be used in order to find the significance and strength contribution of the VRI and the BNP on the goal-function.
Assess the ability of the VRI to aid in classifying the cause of acute dyspnea as HF or COPD | Baseline testing at ED presentation
  The tertiary efficacy analysis set (TEAS) consists of all patients who have final diagnosis (CHF/COPD) & VRI results.
  -Similar to the previous objectives - accuracy (with the GS) and agreement rates (with BNP/NT-proBNP); comparisons based only on CHF and COPD patients.
Evaluate the ability of the VRI to monitor changes in clinical status following treatment in comparison with other standard testing methods (e.g. ECG, serial chest x-rays, etc.) | Baseline testing and repeated testing after 2 hours
  The fourth efficacy analysis set consists of patients who have baseline & after treatment follow-up clinical data & VRI recordings.
  * Descriptive statistics will be used in order to evaluate the changes following treatment in comparison to baseline condition.
  * The changes will be categorized to status of improved, worse or same and will be compared, when available, to existing tools.

CONTACTS AND LOCATIONS:
Overall Officials: Charles V. Pollack, MD, Principal Investigator — Pennsylvania Hospital
Locations (8):
- United States (7):
  - Christiana Care Health System, Newark, Delaware
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Mount Sinai School of Medicine, New York, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - Metrohealth Medical Center, Cleveland, Ohio
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- Beilinson Hospital, Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Wang Z, Bartter T, Baumann BM, Abouzgheib W, Chansky ME, Jean S. Asynchrony between left and right lungs in acute asthma. J Asthma. 2008 Sep;45(7):575-8. doi: 10.1080/02770900802017744. PMID 18773329
- [Background] Guntupalli KK, Reddy RM, Loutfi RH, Alapat PM, Bandi VD, Hanania NA. Evaluation of obstructive lung disease with vibration response imaging. J Asthma. 2008 Dec;45(10):923-30. doi: 10.1080/02770900802395496. PMID 19085584
- [Background] Dellinger RP, Parrillo JE, Kushnir A, Rossi M, Kushnir I. Dynamic visualization of lung sounds with a vibration response device: a case series. Respiration. 2008;75(1):60-72. doi: 10.1159/000103558. Epub 2007 Jun 4. PMID 17551264